CLINICAL TRIAL: NCT00191204
Title: Long Term Monitoring of Safety in Subjects Treated With Duloxetine for Stress Urinary Incontinence
Brief Title: Open Label Phase III Duloxetine Study for Stress Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5309; F1J-MC-SBBM
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Urinary Incontinence Stress
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine

SUMMARY:
The purpose of this study is to monitor the long term safety of duloxetine in the treatment of stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Female out patients
* Are ambulatory and are able to use a toilet independently and without difficulty.

Exclusion Criteria:

* Use of monoamine oxidase inhibitors (MAOIs)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363
Dates: Start 2001-09; Study Completion 2006-05

PRIMARY OUTCOMES:
The primary objective of this study is to generate long-term safety data for duloxetine in the treatment of women with stress urinary incontinence.

SECONDARY OUTCOMES:
The secondary objective of this study is to collect data to demonstrate the maintenance of effect of duloxetine on patients quality of life, measured by Patient Impression of Improvement questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) OR 1-317-615-4559 Mon - Fri 9am - 5pm Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours EST), or speak with your personal physician., Peterborough, United Kingdom